CLINICAL TRIAL: NCT02768259
Title: Prevalence of Pulmonary Arterial Hypertension in Patients With Connective Tissue in Egyptian Patients ( Single Center Study)
Brief Title: Prevalence of Pulmonary Arterial Hypertension in Patients With Connective Tissue Diseases in Egyptian Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Elshazly, Professor of pulmonary Medicine, Cairo University
Other Study IDs: Cairo2000
Record Dates: First submitted 2016-05-08; First posted 2016-05-11 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Connective Tissue Diseases; Pulmonary Hypertension
MeSH Terms: conditions — Connective Tissue Diseases; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
* Measuring the incidence and prevalence of PAH in Egyptian patients with different types of MCD
* Determination of survival & the risk factors of mortality.

DETAILED DESCRIPTION:
PH is defined as a mean pulmonary artery pressure greater than 25 mmHg. PAH can be assessed by different means, however right heart catheterization (RHC) is the gold standard diagnostic method .

Among the different subgroups of pulmonary arterial hypertension (PAH), those associated with connective tissue diseases (CTDs) are a specific entity with distinct hemodynamic and prognostic features reflecting the importance of a rheumatological assessment in PAH, especially with the unfavorable prognostic impact in these patients.

Compared to patients with idiopathic PAH, patients with CTD-associated PAH have a higher mortality and a lower walking distance on the 6-minute walk test, higher levels of B-type natriuretic peptide, worse right ventricular function, more left-sided heart dysfunction, lower lung function, and more pericardial disease.

That's why, PAH screening is routinely performed in systemic sclerosis (SSc) and in other CTDs and also, as suggested by international guidelines, it is important to rule out CTDs in patients with PAH, because patients diagnosed as idiopathic PAH (iPAH) may have an associated CTD previously unrecognized.

Although the similarities in pathogenesis of PAH in CTD such as systemic sclerosis (SSc), systemic lupus erythematosus (SLE), and mixed connective tissue disease (MCTD), there are variabilities in outcomes in patients with CTD-associated PAH.

ELIGIBILITY:
Inclusion Criteria:

- Patients diagnosed as connective tissue diseases fulfilling ACR criteria will be recruited

Exclusion Criteria:

non

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as connective tissue diseases fulfilling ACR criteria will be recruited
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
prevalence | 1 year
  Pulmonary hypertension

SECONDARY OUTCOMES:
Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa I Elshazly, MD, Principal Investigator — Professor of pulmonary Medicine ,Cairo University
Locations (1):
- Kasr Alaini School of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided